CLINICAL TRIAL: NCT03612583
Title: Lung and Diaphragm-Protective Ventilation by Means of Assessing Respiratory Work
Acronym: LANDMARK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-5644
Record Dates: First submitted 2018-07-05; First posted 2018-08-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diaphragm Injury; Lung Injury; Respiratory Insufficiency; Mechanical Ventilation Complication
Keywords: Diaphragm Dysfunction; Acute Respiratory Failure; Sedation; Mechanical Ventilation; Lung Stress
MeSH Terms: conditions — Lung Injury; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower PEEP (Experimental): Lung- and Diaphragm-Protective Ventilation - PEEP will be set at 8 cm H2O
  Interventions: Procedure: Lung- and Diaphragm-Protective Ventilation
- Higher PEEP (Experimental): Lung- and Diaphragm-Protective Ventilation - PEEP will be titrated to achieve end-expiratory PL = 2-3 cm H20 and at least 5 cm H2O greater than the level applied in the lower PEEP arm
  Interventions: Procedure: Lung- and Diaphragm-Protective Ventilation

INTERVENTIONS:
Procedure: Lung- and Diaphragm-Protective Ventilation — Ventilation and sedation will be progressively modified according to the LDPV algorithm to achieve targets. Patients will be crossed-over to the opposite PEEP strategy. LDPV titration will then be repeated to achieve LDPV targets. After establishing a combination of ventilation and sedation settings at which LDPV targets are achieved, the targets will be maintained over a 24-hour period.
  Other Names: LDPV

SUMMARY:
This study is designed to test a proposed strategy for lung- and diaphragm-protective ventilation (LDPV) in patients with acute hypoxemic respiratory failure. Ventilation and sedation will be titrated to evaluate whether it is feasible and safe within this patient population.

DETAILED DESCRIPTION:
Lung injury and diaphragm injury incurred by mechanical ventilation have very serious adverse effects on patients with acute respiratory failure. Lung injury results from excessive mechanical stress and strain applied to the lung by the ventilator and/or respiratory muscles, while diaphragm injury results from either insufficient or excessive inspiratory effort.

The objective of this study is to investigate a new LDPV strategy designed to prevent both disuse-mediated and load-induced diaphragm injury, while also preventing excess global and regional mechanical stress and strain in the injured lung. To achieve these goals, the following specific targets to be met are: (1) respiratory muscle effort similar to that of healthy subjects breathing at rest, (2) lung stress within safe limits, and (3) clinically acceptable gas exchange.

Targets are assessed through measurements of global lung stress, tidal recruitment, inspiratory effort, diaphragm contractile effort and adequacy of respiratory muscle and systemic tissue perfusion. Measurements commence at enrollment and continue for 24 hours consecutively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute hypoxemic respiratory failure
* PaO2:FiO2 ratio less than or equal to 300 mm Hg at time of screening
* Oral endotracheal intubation and mechanical ventilation
* Bilateral airspace opacities on chest radiograph or chest CT scan

Exclusion Criteria:

* Liberation from mechanical ventilation is anticipated within 24 hours
* Intubated for traumatic brain injury or stroke
* Contraindication to esophageal catheterization
* Intracranial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients achieving and maintaining LDPV targets | Assessed after achievement of LDPV targets for 24 hours

SECONDARY OUTCOMES:
Inspiratory effort at lower and higher PEEP levels | Assessed 10 minutes after PEEP and sedation are adjusted
Expiratory diaphragmatic effort at lower and higher PEEP levels | Assessed 10 minutes after PEEP and sedation are adjusted
Lung stress and strain at low and high sweep gas flow rates | Assessed 10 minutes after PEEP and sedation are adjusted
Inspiratory effort at low and high sweep gas flow rates | Assessed 10 minutes after PEEP and sedation are adjusted
Sedative infusion rate at low and high sweep gas flow rates | Assessed 10 minutes after PEEP and sedation are adjusted
Accuracy of artificial intelligence model in predicting patient outcomes | Assessed after completing the 24-hour maintenance period
  We will compare the model's prediction of patient's esophageal pressure, pH and transpulmonary pressure to the actual observed values

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dianti J, Fard S, Wong J, Chan TCY, Del Sorbo L, Fan E, Amato MBP, Granton J, Burry L, Reid WD, Zhang B, Ratano D, Keshavjee S, Slutsky AS, Brochard LJ, Ferguson ND, Goligher EC. Strategies for lung- and diaphragm-protective ventilation in acute hypoxemic respiratory failure: a physiological trial. Crit Care. 2022 Aug 29;26(1):259. doi: 10.1186/s13054-022-04123-9. PMID 36038890